CLINICAL TRIAL: NCT00762216
Title: Rotational Stability of the AcrySof® Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-08-001
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2010-05

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toric (Other): Implantation with the AcrySof® Toric intraocular lens
  Interventions: Device: AcrySof® Toric intraocular lens

INTERVENTIONS:
Device: AcrySof® Toric intraocular lens — Implantation of the AcrySof Toric intraocular lens (IOL) into the eye following cataract extraction surgery

SUMMARY:
To assess the rotational stability and the residual refractive cylinder and patient reported outcomes of the AcrySof Toric intraocular lens after unilateral or bilateral implantation.

ELIGIBILITY:
Inclusion Criteria:

* Monolateral or bilateral cataracts
* anticipated intraocular lens (IOL) power of +10 Diopters (D) ~ +25D
* 0.75 ~ 2.0 D of astigmatism measured preoperatively by Keratometry readings
* able to sign the informed consent, to comply with scheduled visits and other study procedures

Exclusion Criteria:

* Preoperative ocular pathology
* previous intraocular or corneal surgery
* an increased risk for complications which could require vitreoretinal surgery
* corneal irregularities
* corneal opacities
* current contact lens usage
* uncontrolled diabetes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 79 eyes of 71 patients were enrolled into the study. 10 eyes (6 patients) were excluded from analysis for astigmatic keratomy outside of the protocol requirements
Pre-assignment Details: non-randomized
Period: Overall Study
Arm/Group | Toric
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toric
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants] — Age data collected for 69 participants; not provided for 2 participants.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 38
    >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data collected for 69 participants; not provided for 2 participants.
  Participants
    Female | 33
    Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Rotational Stability
Description: Average magnitude of intraocular lens (IOL) rotation from day of surgery to 6-months post-surgery, measured in degrees.
Time Frame: 6 Months post-surgery
Population: 67 eyes (64 patients) were evaluated. Of the original 79 eyes, 10 were excluded from the analysis due to being outside of the protocol specifications. Two (2) additional eyes had no operative intraocular lens (IOL) axis noted on file and were omitted from the analysis of IOL rotation.
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Toric
Number analyzed (Participants) | 67
degrees | 4 (3)

2. Secondary Outcome: Residual Refractive Cylinder
Description: The refractive astigmatism 6 months post-surgery, measured in diopters.
Time Frame: 6 Months post-surgery
Population: 69 eyes (65 patients) were evaluated. Of the original 79 eyes, 10 were excluded from the analysis due to being outside of the protocol specifications.
Measure: Mean (Standard Error); unit: diopters
Arm/Group | Toric
Number analyzed (Participants) | 69
diopters | 0.4 (0.4)

ADVERSE EVENTS:
Description: No adverse events were reported for the 71 patients participating in the study.
Arm/Group | Toric
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No